CLINICAL TRIAL: NCT03305263
Title: Hydroxycloroquin (Plaquenil) Behandling af Gentagne Graviditetstab (Abortus Habitualis) - et Randomiseret, Dobbeltblindet, Placebo Kontrolleret Studium
Brief Title: Hydroxychloroquine (HCQ) for Recurrent Pregnancy Loss
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Henriette Svarre Nielsen, MD, DMSc, Consultant, Head of Recurrent Pregnancy Loss Unit, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCQDenmark; 2016-004981-24 (Other Grant/Funding Number: Regionernes Medicinpulje 15/1719)
Record Dates: First submitted 2017-09-12; First posted 2017-10-09 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Recurrent Pregnancy Loss
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychlorochine HCQ (Experimental): Women in the experimental arm will take 200 mg HCQ tablets every day, starting minimum 2 months (recommended 3-6) prior to conception and continuing until 28 weeks of pregnancy or until the pregnancy is over.
  Interventions: Drug: Hydroxychloroquine
- Hydroxychlorochine HCQ Placebo (Placebo Comparator): Women in the experimental arm will take 200 mg HCQ placebo tablets every day, starting minimum 2 months (recommended 3-6) prior to conception and continuing until 28 weeks of pregnancy or until the pregnancy is over.
  Interventions: Drug: Hydroxychloroquine placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — One tablet a day from inclusion until end of pregnancy or gestational age 28
  Other Names: Placebo
  Arms: Hydroxychlorochine HCQ
Drug: Hydroxychloroquine placebo — One tablet a day from inclusion until end of pregnancy or gestational age 28
  Arms: Hydroxychlorochine HCQ Placebo

SUMMARY:
Recurrent pregnancy loss (RPL) defined as 3 or more pregnancy losses affects approximately 3% of couples trying to achieve parenthood. Most cases of RPL are unexplained and have no effective treatment to improve the chance of a live birth. Exciting indications for using Hydroxychloroquine (HCQ) include: Malaria profylaxis and treatment, systemic and discoid lupus erythematosus (SLE) and rheumatoid athritis (RA). HCQ has been reported to have the following properties (anti-thrombotic, vascular-protective, immunomodulatory, improving glucose tolerance, lipid-lowering, and anti-infectious).

There is no data concerning the benefit of HCQ in RPL. Administration for other indications provides extensive safety data during pregnancy.

This study has the potential to establish support for a new treatment option for unexplained RPL.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 4 confirmed consecutive pregnancy losses prior to gestational age 22+0 in women with unexplained RPL
2. ≥ 3 confirmed consecutive pregnancy losses prior to gestational age 22+0 in women with unexplained RPL with minimum one second trimester loss.

Exclusion Criteria:

1. Age below 18 years or above 39 at inclusion
2. Abnomal uterine anatomi at hysterosalpingography/hysteroscopy or hydrosonography
3. Chromosomal abnormalities within the couple
4. Menstrual cycle below 23 days or above 35 days
5. Lupusantikoagulans positivity or immunoglobulin (Ig)G/IgM anticardiolipinantibodies (≥10 GPL kU/l at Rigshospitalets Laboratorium) or plasma homocystein ≥25 mikrogr./l at repeated measurement with 12 weeks interval.
6. HIV or Hepatitis B or C positive
7. Psoriasis, retinopathy og serious imparied hearing (Contraindications for HCQ)
8. Chronic disease that lead to intake of immunemodulatory drugs or potentially pregnancy toxic agents
9. Hemoglobin ≤ 6.5 mmol/L, leukocytes <3.5 E9/L, platelets <145 E9/L at inclusion
10. Previous treatment with HCQ in pregnancy
11. >1previous live birth
12. previous participation in this trial

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Live birth | At delivery

SECONDARY OUTCOMES:
Live birth after exclusion of patients with a chromosomal abnormal pregnancy loss, extrauterine pregnancy loss, intended abortion or patients with insufficient intake of study medicine | At delivery
Birth weight | At delivery
Gestational age | up to at delivery
Admittance to neonatal unit | Within 28 days of delivery
Immunological status | Up to two years after end of study
  Measuements of celllur and humoral immunity

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided